CLINICAL TRIAL: NCT00898677
Title: A Randomized, Placebo-Controlled, Parallel-Groups, Outpatient Study to Examine the Safety, Tolerability, and Efficacy of Single Oral Doses of MK0462 5 mg, MK0462 10 mg, and Sumatriptan 100 mg for Acute Treatment of Migraine
Brief Title: Rizatriptan 5 mg and 10 mg, Sumatriptan 100 mg, and Placebo Comparison Study (0462-030)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-030; 2009_591
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Results first posted 2009-07-14 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): rizatriptan 5 mg
  Interventions: Drug: rizatriptan benzoate
- 2 (Experimental): rizatriptan 10 mg
  Interventions: Drug: rizatriptan benzoate
- 3 (Active Comparator): sumatriptan 100 mg
  Interventions: Drug: Comparator: sumatriptan
- 4 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: rizatriptan benzoate — single dose administration of 5mg rizatriptan (by Mouth) p.o.
  Other Names: rizatriptan; MK0462
  Arms: 1
Drug: rizatriptan benzoate — single dose administration of 10 mg rizatriptan p.o.
  Other Names: rizatriptan; MK0462
  Arms: 2
Drug: Comparator: sumatriptan — single dose administration of sumatriptan 100 p.o.
  Other Names: sumatriptan
  Arms: 3
Drug: Comparator: Placebo — placebo to rizatriptan
  Arms: 4

SUMMARY:
A study to compare rizatriptan 10 mg verse sumatriptan 100 mg in the treatment of migraine attacks and duration of relief provided. This study will also provide additional efficacy data on rizatriptan 5 mg and 10 mg for the treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patient had at least a 6-month history of migraine, with or without aura
* Patient was male, or if female must have been postmenopausal, surgically sterilized, or taking adequate contraceptive precautions.
* Patient was judged to be in good health, apart from migraine

Exclusion Criteria:

* Patient was pregnant or a nursing mother
* Patient had abused drugs or alcohol within 12 months prior to entering the study
* Patient had a history of cardiovascular disease
* Patient had clinically significant Electrocardiography (ECG) abnormality
* Patient had a resting systolic blood pressure of greater than 145 mm Hg or diastolic of less than 95 mm Hg at screening
* Patient received treatment with an investigational device or compound within 30 days of the study start
* Patient typically suffered from less then 1 or more than 8 attacks of migraine per month
* Patient had difficulty in distinguishing his/her migraine attacks from tension or interval headaches
* Patient had hypersensitivity to sumatriptan
* Patient had participated in any previous study involving rizatriptan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1268 (Actual)
Dates: Start 1995-09; Primary Completion 1996-05 (Actual); Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Ho TW, Rodgers A, Bigal ME. Impact of recent prior opioid use on rizatriptan efficacy. A post hoc pooled analysis. Headache. 2009 Mar;49(3):395-403. doi: 10.1111/j.1526-4610.2009.01346.x. Epub 2008 Feb 12. PMID 19222588
- [Result] Tfelt-Hansen P, Teall J, Rodriguez F, Giacovazzo M, Paz J, Malbecq W, Block GA, Reines SA, Visser WH. Oral rizatriptan versus oral sumatriptan: a direct comparative study in the acute treatment of migraine. Rizatriptan 030 Study Group. Headache. 1998 Nov-Dec;38(10):748-55. doi: 10.1046/j.1526-4610.1998.3810748.x. PMID 11284463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 47 sites in 21 countries in Canada, South America, Europe, Middle East, South Africa, and Australia
  First Patient Treated: September 1995
  Last Patient Treated: May 1996
Pre-assignment Details: Outpatients screened at a pretreatment visit were given allocated drug supply with instructions. If patients had not treated an attack within 2 months of being enrolled, they were required to return for a rescreen visit. If by 4 months after being enrolled patients still had not treated an attack, they were discontinued from the study.
Groups:
- Rizatriptan 5 mg: Rizatriptan 5 mg orally once for treatment of single migraine attack
- Rizatriptan 10 mg: Rizatriptan 10 mg orally once for treatment of single migraine attack
- Sumatriptan 100 mg: Sumatriptan 100 mg orally once for treatment of single migraine attack
- Placebo: Placebo matching Rizatriptan and Sumatriptan orally once for treatment of single migraine attack
Period: Overall Study
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Started | 180 | 455 | 455 | 178
Patients Treated | 164 (Patients Not Treated: 16) | 387 (Patients Not Treated: 68) | 388 (Patients Not Treated: 67) | 160 (Patients Not Treated: 18)
Completed | 163 | 386 | 383 | 159
Not Completed | 17 | 69 | 72 | 19
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Not Treated: Adverse Event | 0 | 2 | 1 | 0
Not completed — Not Treated: Lost to Follow-Up | 0 | 5 | 5 | 2
Not completed — Not Treated: Pregnancy | 0 | 0 | 1 | 0
Not completed — Not Treated: Protocol Violation | 2 | 0 | 2 | 0
Not completed — Not Treated: Withdraw by Subject | 2 | 16 | 11 | 3
Not completed — Not Treated: Patient uncooperative | 2 | 3 | 1 | 0
Not completed — Not Treated: Abnormal Prestudy Labs | 0 | 0 | 0 | 1
Not completed — Not Treated: Abnormal Baseline ECG | 1 | 0 | 0 | 0
Not completed — Not Treated: No Longer Met Inc Criteria | 0 | 3 | 1 | 0
Not completed — Not Treated: Lack of Migraine Attack | 9 | 39 | 43 | 12
Not completed — Not Treated: Other (Not Specified) | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rizatriptan 5 mg: Rizatriptan 5 mg orally once for treatment of single migraine attack.
  Baseline measure Participants reported are those participants that recieved study treatment.
- Rizatriptan 10 mg: Rizatriptan 10 mg orally once for treatment of single migraine attack
  Baseline measure Participants reported are those participants that recieved study treatment.
- Sumatriptan 100 mg: Sumatriptan 100 mg orally once for treatment of single migraine attack
  Baseline measure Participants reported are those participants that recieved study treatment.
- Placebo: Placebo matching Rizatriptan and Sumatriptan orally once for treatment of single migraine attack
  Baseline measure Participants reported are those participants that recieved study treatment.
- Total: Total of all reporting groups
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo | Total
Number analyzed (Participants) | 164 | 387 | 388 | 160 | 1099
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.3) | 37.0 (10.0) | 39.2 (10.1) | 38.3 (10.3) | 38.2 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 319 | 309 | 132 | 898
  Male | 26 | 68 | 79 | 28 | 201
Baseline Headache Severity [Number; unit: participants] — Each patient rated headache severity on a 4-grade scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain).
  participants
    Grades 1, 0: Mild, no pain, or missing | 0 | 0 | 1 | 1 | 2
    Grade 2: Moderate | 72 | 174 | 191 | 75 | 512
    Grade 3: Severe | 92 | 213 | 196 | 84 | 585
Race/Ethnicity [Number; unit: participants]
  Caucasian | 117 | 282 | 281 | 120 | 800
  Black | 1 | 5 | 3 | 0 | 9
  Asian | 0 | 1 | 2 | 0 | 3
  Hispanic | 33 | 80 | 77 | 32 | 222
  Mestizo | 9 | 15 | 22 | 7 | 53
  Mexican | 0 | 2 | 2 | 0 | 4
  Colored | 0 | 0 | 1 | 0 | 1
  Mexican/Hispanic | 1 | 0 | 0 | 0 | 1
  Mixed | 2 | 2 | 0 | 1 | 5
  Asian/Caucasian | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at 2 Hours After Dose
Description: Patients reporting pain relief defined as a reduction of headache severity from grades 2 or 3 (moderate or severe pain) at baseline to grades 0 or 1 (no headache or mild pain) at 2 hours after treatment
Time Frame: 2 hours after dose
Population: An "all-patients-treated" approach was used in the primary analysis, including all patients who had at least one assessment of pain severity within 2 hours after test medication. Missing values in the treatment phase (i.e., after the baseline phase) were imputed by carrying forward the preceding values in the same phase.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Number analyzed (Participants) | 164 | 385 | 387 | 159
Participants
  2-hour pain relief | 99 | 258 | 239 | 64
  No 2-hour pain relief | 65 | 127 | 148 | 95

2. Primary Outcome: Time to Relief Within 2 Hours After Dose
Description: Patients reporting time to relief defined as the first time point at which a patient reported headache severity grade 1 or 0 (mild pain or no headache) within 2 hours after dose
Time Frame: within 2 hours after dose
Population: An "all-patients-treated" approach was used in the primary analysis, including all patients who had at least one assessment of pain severity within 2 hours after test medication.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Number analyzed (Participants) | 164 | 385 | 387 | 159
Participants
  First pain relief within 2 hrs | 102 | 265 | 247 | 72
  Pain relief did not occur within 2 hrs | 62 | 120 | 140 | 87

3. Secondary Outcome: Pain Free at 2 Hours After Dose
Description: Patients pain free (defined as a reduction of headache severity to grade 0 [no pain]) at 2 hours after treatment. Each patient rated headache severity on a 4-point scale (0 = no headache; 1 = mild pain; 2 = moderate pain; 3 = severe pain).
Time Frame: 2 hours after dose
Population: An "all-patients-treated" approach was used in the secondary analysis, including all patients who had at least one assessment of pain severity within 2 hours after test medication. Missing values in the treatment phase (i.e., after the baseline phase) were imputed by carrying forward the preceding values in the same phase.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Number analyzed (Participants) | 164 | 385 | 387 | 159
Participants
  2-hour Pain freedom | 41 | 155 | 127 | 15
  No 2-hour pain freedom | 123 | 230 | 260 | 139

4. Secondary Outcome: Functional Status at 2 Hours After Dose
Description: Patients with no functional disability measured by the level of impairment to daily activities at 2 hours after treatment. Each patient rated functional disability on a 4-grade scale (0 = no functional disability; 1 = daily activities mildly impaired; 2 = daily activities severely impaired; 3 = unable to carry out daily activities, requires bed rest).
Time Frame: 2 hours after dose
Population: An "all-patients-treated" approach was used in the secondary analysis. Missing data were replaced by carrying forward the preceding value.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Number analyzed (Participants) | 164 | 385 | 387 | 159
Participants
  No functional disability | 52 | 160 | 126 | 31
  Mildly impaired | 62 | 123 | 142 | 59
  Severely impaired | 27 | 60 | 67 | 33
  Required bed rest | 23 | 42 | 52 | 36

5. Secondary Outcome: Nausea at 2 Hours After Dose
Description: Patients who recorded the presence or absence of nausea 2 hours after dose
Time Frame: 2 hours after dose
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Number analyzed (Participants) | 164 | 385 | 387 | 159
participants
  2-hour Nausea | 37 | 95 | 128 | 68
  No 2-hour Nausea | 127 | 290 | 259 | 91

ADVERSE EVENTS:
Time Frame: During the 24 hours treatment period, and up to and including 7 days after the last dose of study therapy.
Description: Although a patient may have had two or more adverse experiences the patient is counted only once in a category. The same patient may appear in different categories.
  Adverse Event participants reported are those participants that received study treatment and had safety follow-up.
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Sumatriptan 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/164 | 0/387 | 0/388 | 0/160
Other Adverse Events (participants affected / at risk) | 62/164 | 159/387 | 188/388 | 51/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=164) | Rizatriptan 10 mg (N=387) | Sumatriptan 100 mg (N=388) | Placebo (N=160)
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 5 mg (N=164) | Rizatriptan 10 mg (N=387) | Sumatriptan 100 mg (N=388) | Placebo (N=160)
Asthenia/Fatigue (General disorders) | 4 | 30 | 32 | 6
Chills (General disorders) | 3 | 3 | 6 | 1
Cold Sensation (General disorders) | 2 | 4 | 4 | 4
Fever (General disorders) | 1 | 2 | 2 | 2
Pain, Abdominal (General disorders) | 7 | 12 | 20 | 2
Pain, Chest (General disorders) | 2 | 13 | 22 | 4
Warm Sensation (General disorders) | 2 | 2 | 0 | 1
Palpitation (Cardiac disorders) | 7 | 6 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 3 | 7 | 2
Acid Regurgitation (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 3 | 1
Dry Mouth (Gastrointestinal disorders) | 4 | 9 | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 6 | 1
Nausea (Gastrointestinal disorders) | 8 | 22 | 35 | 4
Vomiting (Gastrointestinal disorders) | 5 | 12 | 10 | 8
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Alanine Aminotransferase Increased (Metabolism and nutrition disorders) | 2 | 2 | 3 | 1
Aspartate Aminotransferase Increased (Metabolism and nutrition disorders) | 3 | 1 | 5 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Heaviness, Regional (Musculoskeletal and connective tissue disorders) | 1 | 10 | 9 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 0
Pain, Neck (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 2
Pain, Shoulder (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 9 | 1
Depression (Psychiatric disorders) | 3 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 9 | 30 | 35 | 6
Headache (Nervous system disorders) | 3 | 12 | 11 | 2
Hypesthesia (Nervous system disorders) | 1 | 2 | 9 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 6 | 2
Nervousness (Psychiatric disorders) | 1 | 1 | 4 | 0
Paresthesia (Nervous system disorders) | 3 | 11 | 16 | 5
Somnolence (Psychiatric disorders) | 13 | 32 | 28 | 9
Tremor (Nervous system disorders) | 4 | 1 | 8 | 1
Discomfort, Pharyngeal (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 11 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4 | 1
Flushing (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 1
Sweating (Skin and subcutaneous tissue disorders) | 1 | 5 | 10 | 1
Blurred Vision (Eye disorders) | 0 | 3 | 5 | 0
Perversion, Taste (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Hot Flashes (Reproductive system and breast disorders) | 1 | 4 | 8 | 2
Urinary Frequency (Renal and urinary disorders) | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.